CLINICAL TRIAL: NCT01641965
Title: Impact of Early Non-invasive Ventilation in Amyotrophic Lateral Sclerosis Patients: a Randomized Controlled Trial
Brief Title: Impact of Early Non Invasive Ventilation in Amyotrophic Lateral Sclerosis (ALS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Eva Farrero Munoz, Medical Doctor, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC 111/11
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early non invasive ventilation (Active Comparator): Patients assigned to this arm will start non invasive ventilation with home pressure ventilator model Vivo 40 (BREAS Medical AB)immediately after randomization (when their FVC reaches the threshold of the 75% of the predicted value)
  Interventions: Device: Home pressure ventilator model Vivo 40 (BREAS Medical AB)
- standard (Active Comparator): patients in this arm will start non invasive ventilation with home pressure ventilator model Vivo 40 (BREAS Medical AB) when they fulfil at least one of the following criteria: (i) FVC < 50% predicted, (ii) orthopnea, and/or (iii) PaCO2 > 45 mmHg.
  Interventions: Device: Home pressure ventilator model Vivo 40 (BREAS Medical AB)

INTERVENTIONS:
Device: Home pressure ventilator model Vivo 40 (BREAS Medical AB) — Nocturnal non invasive ventilation (Vivo 40)with minimum pressure support of 10 cm H2O (IPAP 14, EPAP 4). Parameters will be adjusted according to tolerance and to achieve PaCO2 < 45 mmHg and improve symptoms.

SUMMARY:
Timing of initiating domiciliary no invasive ventilation (NIV) in amyotrophic lateral sclerosis patients remains unclear. The hypothesis of the study is that the early use of NIV, in the initial phase of respiratory muscle weakness, improves the prognosis of ALS patients.

Principal objective: To evaluate the impact of early NIV in the survival of ALS patients.

Secondary objectives:To determine the effects from early NIV in the progression of respiratory muscle weakness. To analyze the impact of early NIV in the quality of life of ALS patients. To evaluate the correlation between the FVC and other parameters of respiratory evaluation (maximal inspiratory pressure (MIP), sniff nasal inspiratory pressure (SNP), nocturnal desaturation) and their utility in the early indication of the NIV. To evaluate the tolerance to the early NIV.

Methods: multicentric, randomized, open-label, controlled clinical trial with a parallel treatment design. Patients will be included when their FVC reaches the threshold of the 75% of the predicted value and will be randomized in: Group A: the NIV treatment will begin immediately and Group B: the NIV treatment will be started when patients fulfil at least one of the following criteria: (i) FVC < 50% predicted, (ii) orthopnea, and/or (iii) PaCO2 > 45 mmHg. Follow-up visits will be done every three months with pulmonary function test, nocturnal pulse oximetry, quality of life and quality of sleep tests, assessment of disease progression (ALSFSR-R scale), tolerance and compliance with NIV.

DETAILED DESCRIPTION:
ALS patients with early impairment of respiratory muscles (FVC around 75%) will be radomised to initiate NIV or conventional follow-up.

The NIV treatment will be initiated during a hospital with the model of ventilator VIVO 40 (BREAS Medical AD, Sweden) using a pressure support assisted/control mode, with a minimum pressure support 10 cm.

Initial NIV indication in both groups of patients will nocturnal. Patients will be defined as tolerant to NIV if they do not refer inconveniences and is able to asleep with NIV.

The efficacy of the intervention will be compared in both groups with survival until death or change to invasive tracheal ventilation as a prymary efficacy parameter.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Definite ALS diagnosis according to El Escorial Criteria
* Ability to understand and perform the pulmonary function test
* FVC ≤ 75% (with FVC registry >75% documented within the six previous months)

Exclusion Criteria:

* Major comorbidity (non-related with ALS) that can shorten life expectancy
* Cognitive impairment that prevents the patient to understand and perform the study procedures including technically acceptable pulmonary function tests (FVC, MIP, SNP, PCF)
* Patient refusal of NIV treatment
* Previous respiratory or cardiac diseases with known impaired spirometry
* Indication of NIV according to standard criteria (PaCO2 > 45 mmHg, FVC < 50%, orthopnea)
* ALS with slow disease progression (more than 3 years)
* Participation in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
survival until death or tracheostomy | three years
  To evaluate the impact of the early use of NIV in the survival function of the time until death or tracheostomy of ALS patients, compared with a standard initiation of NIV.

SECONDARY OUTCOMES:
effects from early use of NIV in progression of respiratory muscle weakness | three years
  To determine the effects from early use of NIV in progression of respiratory muscle weakness, measured by rate of decline in FVC

CONTACTS AND LOCATIONS:
Overall Officials: Eva Farrero, MD, Principal Investigator — Hospital Universitari Bellvitge
Locations (1):
- Hospital Universitari Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarasate M, Gonzalez N, Cordoba-Izquierdo A, Prats E, Gonzalez-Moro JMR, Marti S, Lujan M, Calle M, Anton A, Povedano M, Farrero E. Impact of Early Non-Invasive Ventilation in Amyotrophic Lateral Sclerosis: A multicenter Randomized Controlled Trial. J Neuromuscul Dis. 2023;10(4):627-637. doi: 10.3233/JND-221658. PMID 37212068